CLINICAL TRIAL: NCT05452668
Title: Effectiveness of Laser Therapy of Different Wavelengths in Chemotherapy Induced Oral Mucositis in Children With Acute Lymphoblastic Leukemia
Brief Title: Laser Therapy Effect on Oral Mucositis in Childhood Acute Lymphoblastic Leukemia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CCHE-ALL004
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Oral Mucositis; Childhood Acute Lymphoblastic Leukemia
Keywords: Oral Mucositis; Childhood Acute Lymphoblastic Leukemia; Laser therapy; low level laser therapy
MeSH Terms: conditions — Stomatitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome evaluator will be a single personnel from the oncology team following up with the case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Seventeen patients will receive treatment using the red wavelength (660 nm) to provide biostimulation. Plus the current protocol (antifungal +/- antiviral and analgesics) used by CCHE which will be recorded in the patient's file.
  Interventions: Device: Laser Therapy
- Group II (Experimental): Seventeen patients will receive treatment using the infrared wavelength (970 nm) to provide biosstimulation. plus the current protocol(antifungal +/- antiviral and analgesics) used by CCHE which will be recorded in the patient's file.
  Interventions: Device: Laser Therapy
- Group III (Sham Comparator): Seventeen patients will receive mock treatment which is the exact repetition of the treatment modality but without any laser emission plus the current protocol(antifungal +/- antiviral and analgesics) used by CCHE which will be recorded in the patient's file
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: Laser Therapy — - Laser will be applied with the specified wave length using a diode laser device over 4 consecutive days.
  Arms: Group I; Group II
Device: Sham procedure — Seventeen patients will receive mock treatment which is the exact repetition of the treatment modality but without any laser emission plus the current Protocol(antifungal +/- antiviral and analgesics) used by CCHE which will be recorded in the patient's file
  Arms: Group III

SUMMARY:
Introduction: Oral mucositis is one of the most frequent complications associated with chemotherapy, occurring in up to 90% children receiving treatment for cancer. Different treatment modalities have been suggested with inconsistent results. Recently, it has been suggested that the use of laser could reduce the grade of oral mucositis and alleviate the symptoms.

Aim: To evaluate and compare the efficacy between the high (Infrared) wavelength laser and low (red) wavelength laser in management of chemotherapy induced oral mucositis in children with acute lymphoblastic leukemia.

Methods: This study is a randomized, prospective, double-blind trial that will include acute lymphoblastic leukemia inpatients receiving induction chemotherapy between the age of 3 and 14years who develop oral mucositis grade 2 or more. These patients will be randomized by the Clinical Epidemiology unit using a computer-based method into three groups. Group I: will be treated with Laser wavelength 660 nm, group II: will be treated with laser wavelength 970 nm, and group III: will receive mock treatment which is the exact repetition of the treatment modality but without any laser emission. All the patients will follow the hospital standard management for oral mucositis. All patients will be assessed for pain score using CHIMES, oral mucositis using NCI-CTCAE scale V5 on days, 0,4,7 and 11. As well as measuring the duration of the lesion.

DETAILED DESCRIPTION:
This study is a randomized, prospective, double-blind trial that will include acute lymphoblastic leukemia inpatients receiving induction chemotherapy between the age of 3 and 14 years who develop oral mucositis grade 2 or more. These patients will be randomized by the Clinical Epidemiology unit using a computer-based method into three groups.

Group I: will be treated with Laser wavelength 660 nm, Group II: will be treated with laser wavelength 970 nm, Group III: will receive mock treatment which is the exact repetition of the treatment modality but without any laser emission.

All the patients will follow the hospital standard management for oral mucositis.

All patients will be assessed for

1. Pain score using CHIMES,
2. Oral mucositis using NCI-CTCAE scale V5 on days, 0,4,7 and 11.
3. Measuring the duration of the lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Acute Lymphoblastic Leukemia in the induction therapy phase and have oral mucositis grade 2 or more.
2. Age: 3-14 years old of both genders.
3. No previous treatment with laser.
4. Ability to open mouth for more than 2 cm for the duration of laser application with a level of cooperation (Frankl rating 3 or 4).
5. Patients who still have 10 days in their induction therapy phase or can be followed up for a mininum of 10 days after the development of oral mucositis

Exclusion Criteria:

1. Patients receiving radiotherapy
2. Received oral Cryotherapy or IV keratinocyte growth factor for oral mucositis
3. Patients with unstable clinical condition (e.g. sepsis)
4. Patients who will be withdrawn from participation according to their request or due to loss in follow up

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | 4 days
  Assessing the change from baseline pain at day 4. Pain assessment will be done by Children's International Mucositis Evaluation Scale (ChIMES).
  For children less than 8 years the guardian will assist the child in filling the chart. Pain will be measured on day 0, 4, 7 and 11

SECONDARY OUTCOMES:
Oral Mucositis Severity: | 4 days
  Assessing the change in the Oral Mucositis Severity from baseline at day 4. his will be measured using the National Cancer Institute Common Toxicity Criteria for adverse events (NCI-CTCAE) scale version 5

CONTACTS AND LOCATIONS:
Overall Officials: Hussein ElNoury, MSc, Principal Investigator — NewGiza University
Locations (2):
- Egypt (2):
  - Children Cancer Hospital Egypt 57357, Cairo
  - Children Cancer Hospital in Egypt 57357, Cairo

IPD SHARING:
Plan to Share IPD: No